CLINICAL TRIAL: NCT01475890
Title: Safe and Effective Vitamin D Supplementation in HIV
Brief Title: Vitamin D Supplementation in HIV
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-008093; 5R01AT005531-02 (NIH)
Record Dates: First submitted 2011-09-13; First posted 2011-11-22 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: HIV-infection/Aids
Keywords: HIV/AIDS; Nutrition
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7000IU/day (Active Comparator): 29 subjects will be randomized to receive 7000IU/day of vitamin D3.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): 29 subjects will be randomized to receive placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 7000IU per day of vitamin D3 for 12 months.
  Arms: 7000IU/day
Dietary Supplement: Placebo — Once a day for 12 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of vitamin D supplementation in children, adolescents and young adults with Human Immunodeficiency Virus and acquired immunodeficiency syndrome (HIV/AIDS). The study is a 12-month randomized, double blind, placebo-controlled study of vitamin D3 (vit D) supplementation using 7000IU/day based on evidence from the Vit D Dose Finding Study-IRB 09-007332.

DETAILED DESCRIPTION:
Optimal vitamin D (vit D) concentration and metabolism are essential for normal immune function, growth, muscle, bone, and inflammatory status in children, adolescents and adults with HIV/AIDS. The impact of vit D supplementation will be evaluated for safety and efficacy using clinically important outcomes, and this will overcome the critical barrier for use of vit D supplementation in research and clinical care. Inexpensive and easy to administer, vit D supplementation may prove to be an effective and feasible treatment for symptoms and prevention of side effects for people of all ages living with HIV/AIDS in the US and around the world.

The study is a 12-month randomized, double blind, placebo-controlled study of vitamin D3 (vit D) supplementation using 7000IU/day based on evidence from the Vit D Dose Finding Study-IRB 09-007332 in 58 subjects with both Perinatally Acquired (PA) and Behaviorally Acquired (BA) HIV/AIDS to assess the long-term safety in terms of serum calcium and 25OHD concentrations, and efficacy in terms of the effect of vit D supplementation on 25OHD, cathelicidin, growth (pre- and peripubertal participants), body composition, bone, muscle, immune and inflammatory status and HIV/AIDS disease severity and progression.

Primary Hypotheses:

H1: Vit D supplementation is safe and does not result in an increased incidence of elevated serum calcium (above age-specific range) associated with elevated serum 25OHD (>160 ng/mL) in treated subjects compared with the subjects receiving placebo.

H2: Vit D supplementation is significantly associated with both increased 25D and cathelicidin in treated subjects compared with subjects receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

1. HIV seropositive diagnosed with standard techniques
2. Age for PA Group: 5.0 to 24.9 y
3. Age for BA Group: 15.0 to 24.9 y
4. In usual state of good health (no hospitalizations, emergency room or unscheduled acute illness visits for 2 weeks prior to enrollment)
5. Subject and/or family commitment to the 12-month study

Exclusion Criteria:

1. Other chronic health conditions that may affect growth, dietary intake, and/or nutritional status
2. Pregnancy
3. Participation in another HIV intervention study with impact on 25D serum concentrations
4. Use of vit D3 supplementation for the purpose of treating vit D deficiency
5. Use of vit D3 supplementation not part of a prescribed treatment plan for vit D deficiency (subjects willing to discontinue supplementation will become eligible after a minimum of a 2 month washout period)
6. Non-English Speaking

Ages: 5 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Vitamin D Supplementation Safety | 12 months
  elevated serum calcium (above age-specific range) associated with elevated serum 25D (>160 ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia A Stallings, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Rovner AJ, Stallings VA, Rutstein R, Schall JI, Leonard MB, Zemel BS. Effect of high-dose cholecalciferol (vitamin D3) on bone and body composition in children and young adults with HIV infection: a randomized, double-blind, placebo-controlled trial. Osteoporos Int. 2017 Jan;28(1):201-209. doi: 10.1007/s00198-016-3826-x. Epub 2016 Nov 11. PMID 27837268
- [Derived] Brown JC, Schall JI, Rutstein RM, Leonard MB, Zemel BS, Stallings VA. The impact of vitamin D3 supplementation on muscle function among HIV-infected children and young adults: a randomized controlled trial. J Musculoskelet Neuronal Interact. 2015 Jun;15(2):145-53. PMID 26032206